CLINICAL TRIAL: NCT01434329
Title: S8600-S9031-S9333-A, Identification of Differentially Methylated Genomic Regions That Are Prognostically Significant in AML
Brief Title: S8600-S9031-S9333-A, Study of DNA in Samples From Patients With Acute Myeloid Leukemia
Status: Completed | Type: Observational
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: S8600-S9031-S9333-A; S8600-S9031-S9333-A (Other: SWOG); U10CA032102 (NIH)
Record Dates: First submitted 2011-09-13; First posted 2011-09-14 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Leukemia
Keywords: untreated adult acute myeloid leukemia
MeSH Terms: conditions — Leukemia | interventions — DNA Methylation; Gene Expression Profiling; Microarray Analysis

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: DNA methylation analysis
Genetic: gene expression analysis
Genetic: microarray analysis
Other: laboratory biomarker analysis
Other: medical chart review

SUMMARY:
RATIONALE: Studying samples of blood and bone marrow from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors predict how patients respond to treatment.

PURPOSE: This research trial studies DNA in samples from patients with acute myeloid leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* To identify differentially methylated regions (DMRs) associated with overall survival (OS) of acute myeloid leukemia (AML) patients with normal cytogenetics.
* To develop and evaluate in an independent validation set a prognostic score for OS based on the identified DMR.
* To determine whether the prognostic score can group patients into risk groups based on OS.

OUTLINE: Archived blood or bone marrow samples are analyzed for DNA methylation alterations by CHARM array-based genome assay. Each patient's clinical data is also collected.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* De novo acute myeloid leukemia (AML) patients with normal cytogenetics treated with curative therapy who survived at least 28 days after therapy started
* Samples will be taken from the following studies: SWOG-8600, SWOG-9031, SWOG-9333, SWOG-9500, SWOG-S9918, SWOG-S0106, and SWOG-S0112

  * Blood or marrow specimens can be used

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients enrolled on S8600, S9031 or S9333 who consented to use of specimens for future research
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2011-10; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Identification of DMRs associated with OS | immediate
Development and evaluation of a prognostic score of OS based on DMRs identified | immediate
Prognostic score able to group AML patients into risk groups | immediate

CONTACTS AND LOCATIONS:
Overall Officials: Min Fang, MD, PhD, Principal Investigator — Fred Hutchinson Cancer Center